CLINICAL TRIAL: NCT00416559
Title: Phase II Trial of Surgery as the Only Treatment for INSS Stage 2A & 2B Neuroblastoma
Brief Title: Observation of Young Patients With Localized Neuroblastoma Who Have Undergone Surgery Only
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Supportive Care
Other Study IDs: CDR0000454574; CCLG-NB-1995-06; EU-20596; CCLG-94-01
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2007-05

CONDITIONS: Long-term Effects Secondary to Cancer Therapy in Children; Neuroblastoma
Keywords: long-term effects secondary to cancer therapy in children; localized resectable neuroblastoma; localized unresectable neuroblastoma; regional neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Watchful Waiting

INTERVENTIONS:
Other: clinical observation

SUMMARY:
RATIONALE: Observation is closely monitoring a patient's condition and not giving treatment until symptoms appear or change. Observation may help doctors see how effective surgery is in treating neuroblastoma.

PURPOSE: This phase II trial is studying how well surgery alone works in treating young patients with localized neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the safety and efficacy of surgical treatment alone in young patients with stage 2 neuroblastoma without N-myc amplification (NMA).

Secondary

* Determine predictive factors of relapse and survival of patients with stage 1, 2A, or 2B neuroblastoma without NMA who have undergone surgery only.

OUTLINE: This is a nonrandomized, multicenter study.

Patients with stage 1 or 2 disease and no N-myc amplification (NMA) undergo observation comprising clinical evaluation, ultrasound or CT scan of the abdomen, and chest x-ray periodically for up to 5 years. All other patients undergo additional therapy and follow-up according to national standards. Patients who develop recurrent disease or disease progression may undergo surgical resection, preceded or followed by chemotherapy, according to national standards.

PROJECTED ACCRUAL: A total of 140 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed neuroblastoma or ganglioneuroblastoma
* Meets 1 of the following International Neuroblastoma Staging System (INSS) criteria:

  * Stage 1
  * Stage 2A or 2B meeting 1 of the following criteria:

    * With or without N-myc amplification
    * No evaluation of NMA
    * Symptomatic spinal cord compression
  * Stage 3*
  * Dumbbell syndrome with clinical signs of spinal cord compression*
* NOTE: *These patients are eligible for the study but do not undergo observation; instead they will undergo standard treatment
* Has undergone complete or gross surgical resection OR diagnostic surgical or needle biopsy
* No metastases within 1 month of diagnosis

  * No skin metastases by clinical examination and MIBG scan
  * Normal liver by CT scan or ultrasonography
  * Normal chest X-ray (in case of nonthoracic primary site)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior steroids allowed
* No prior chemotherapy

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Estimated)
Dates: Start 2004-12

PRIMARY OUTCOMES:
Safety and efficacy

SECONDARY OUTCOMES:
Predictive factors of relapse and survival

CONTACTS AND LOCATIONS:
Overall Officials: Bruno De Bernardi, MD, Study Chair — Istituto Giannina Gaslini; Jean Marie Michon, MD — Institut Curie